CLINICAL TRIAL: NCT05796401
Title: PsyCARE Trial - "Efficiency of a Composite Personalised Care on Functional Outcome in Early Psychosis : A Prospective Randomised Controlled Trial "
Brief Title: Efficiency of a Composite Personalised Care on Functional Outcome in Early Psychosis
Acronym: PSYCARE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: D22-P006
Record Dates: First submitted 2023-03-16; First posted 2023-04-03 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-03

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Cognitive Training; Leucovorin; Docosahexaenoic Acids; Therapeutics

STUDY DESIGN:
Intervention Model Description: Phase III, Prospective Randomised Open, Blinded End-point (PROBE) controlled trial stratified according to the developmental burden and centre, with 2x2 factorial designs (equivalent to a 4-arms clinical trial) in a 1:1:1:1 ratio.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment as usual (TAU) (Active Comparator)
  Interventions: Other: Treatment as usual (TAU)
- TAU + cognitive training (Experimental)
  Interventions: Behavioral: Cognitive training; Other: Treatment as usual (TAU)
- TAU + personalized neuroprotective strategies (Experimental)
  Interventions: Drug: Personalized neuroprotective strategies : Vitamin B12, folinic acid, Omega 3, NAC; Other: Treatment as usual (TAU)
- TAU + personalized neuroprotective strategies + cognitive training (Experimental)
  Interventions: Behavioral: Cognitive training; Drug: Personalized neuroprotective strategies : Vitamin B12, folinic acid, Omega 3, NAC; Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Cognitive training — Cognitive reinforcement using digital applications (PSYCARE application) during 12 weeks
  +/- virtual reality based cognitive remediation application : 24 sessions over 12 weeks (only for patients who have a higher cognitive deficits (TMTB score >110s))
  Arms: TAU + cognitive training; TAU + personalized neuroprotective strategies + cognitive training
Drug: Personalized neuroprotective strategies : Vitamin B12, folinic acid, Omega 3, NAC — Personalised neuroprotective medication adapted to the individual's biological profile :
  * Vitamin B12 : 500 micrograms per day
  * Folinic acid : 50 mg per day
  * Omega 3 : 1380 mg EicosaPentaenoic Acid (EPA) + 1140 mg DocosaHexaenoic Acid (DHA) per day
  * N-acetyl-cysteine (NAC) : 2400 mg per day
  duration of supplementation(s) : 12 weeks
  Arms: TAU + personalized neuroprotective strategies; TAU + personalized neuroprotective strategies + cognitive training
Other: Treatment as usual (TAU) — Treatment as usual (TAU), including a standardised psycho-education program with a group cognitive behavioural therapy (e.g. I_Care - You Care) and, in FEP only, second generation antipsychotic from a restricted list (following the recommendations www.orygen.org.au)

SUMMARY:
Chronic psychosis, including schizophrenia is now viewed as a progressive disorder where cognitive deficits predate the clinical onset. Early intervention programs improve the general outcome with staged care strategies, supporting the view that the period before and around the first episode of psychosis is a window of opportunity for improving its functional recovery.

Pioneering epigenetic analyses indicate that psychosis onset involves oxidative stress and inflammation suggesting that neuroprotective strategies could limit or even prevent the onset of or the transition into a chronic disorder. Several biological factors associated with the emergence of psychosis can all be rectified by using safe and easily accepted supplements including alterations folate deficiency/hyperhomocysteinemia; redox imbalance and deficit in polyunsaturated fatty acids (PUFA). The prevalence of these anomalies (20-30%) justifies a systematic detection and could guide personalised add-on strategy.

Cognitive remediation improves quality of life (QoL) and functional outcome in patients with chronic psychosis. It would even be more efficacious in the early phase of psychosis by tackling the negative impact of psychosis on education achievement and employment. However, cognitive dysfunctions are often overlooked in patients at ultra-high risk (UHR) for psychosis and patient with a first episode of psychosis (FEP) and cognitive remediation is not always accessible. New technologies can provide us with youth-friendly, non-stigmatising tools, such as applications with cognitive strategies, motivational tools and functioning guidance personalised according to the need of each individual. Patients can have access to it, wherever they live.

Early psychosis can be associated with inflammation, metabolic deficiency, as well as early structural brain anomalies that reflect brain plasticity abilities and could influence the prognosis and response to cognitive training.

The study hypothesis is that promoting neuroplasticity by cognitive training and personalised virtual psychoeducation guidance could attenuate or reverse early cognitive deficits and improve the overall functional outcome in young patients UHR or FEP and that this effect is modulated by individual brain plasticity abilities. The overall objective of PsyCARE_trial is to improve early intervention in psychosis by providing a composite personalised care (CPC) that will enable personalised cognitive training and psychoeducation guidance, adapted to individuals' needs, cognitive abilities and biological background.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent and young adults, both sexes, aged 15 to 30 years,
* From Community or academic clinics,
* Characterised as UHR or FEP according to the first four items of the Comprehensive Assessment of At Risk Mental State (CAARMS) (first subscale for psychosis) [8] during the last 12 months,
* Informed and written signed consent,
* Participant with regular health insurance

Exclusion Criteria:

* Severe and unstabilised medical conditions,
* Insufficient level in reading and/or French language,
* Current participation in another intervention trial,
* Enforced hospitalization ,
* Intellectual Deficiency (i.e. Intelligence Quotient<70), and / or sensorimotor deficits incompatible with the cognitive training,
* Former treated episode of psychosis, chronic schizophrenia, schizoaffective, or Bipolar disorder,
* Current severe depression (i.e. MADRS > 34),
* Receiving therapeutic levels of antipsychotics for more than 12 months,
* Current medication with benzodiazepine >30 mg per day equivalent diazepam
* Current daily use of substance of abuse (higher than an average equivalent of daily number of 5 cannabis cigarettes). Current severe substance use disorder except for nicotine (SUD, Diagnostic and Statistical Manual of Mental Disorders version V (DSMV criteria) during the last 6 months and/or former severe SUD or dependence DSMIV during more than 5 years.
* Current cognitive remediation programme,
* Pregnant women, parturients, and lactating women,
* Individuals deprived of their liberty by a judicial or administrative decision,
* Individuals of legal age who are the subject of a legal protection measure or unable to express their consent

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Global functioning | 3 to 4 months after the beginning of intervention
  Global functioning will be assessed using the Personal and Social Performance Scale (PSP), a well-validated tool for the measurement of social functioning previously used in early psychosis.
  PSP is a 100-point single-item rating scale (minimum value 1; maximum value: 100). The scale evaluates four main areas: 1) socially useful activities; 2) personal and social relationships; 3) self-care; and 4) disturbing and aggressive behaviours during a determined reference period

SECONDARY OUTCOMES:
Persistence of efficacy on global functioning | 6 to 8 months after the beginning of intervention
  Score on the Personal and Social Performance Scale (PSP)
  PSP is a 100-point single-item rating scale (minimum value 1; maximum value: 100). The scale evaluates four main areas: 1) socially useful activities; 2) personal and social relationships; 3) self-care; and 4) disturbing and aggressive behaviours during a determined reference period
Persistence of efficacy on global functioning | at baseline, then 3 to 4 months and 6 to 8 months after the beginning of intervention
  Scores at Global Functioning Scale-Social and Role [120], measured at V2 and V3. This scale provides a 1 to 10 score separately for social role and for functioning.
Efficiency of Composite Personalised Care (CPC) on clinical outcome (1) | at baseline, then 3 to 4 months and 6 to 8 months after the beginning of intervention
  Comprehensive Assessment of At Risk Mental State (CAARMS) CAARMS evaluates seven dimensions of symptomatology. It provides operational criteria to categorise subjects as 'at-risk' or as psychotic (psychosis threshold) on the basis of the first subscale (10 min), 'positive symptoms' encompassing four sub-scales (Unusual Thought Content, Non-Bizarre Ideas, Perceptual Abnormalities, Disorganised Speech)
Efficiency of Composite Personalised Care (CPC) on clinical outcome (2) | at baseline, then 3 to 4 months and 6 to 8 months after the beginning of intervention
  - SOFAS (Social and Occupational Functioning Assessment Scale or EFSP. SOFAS specifically estimates social functioning on a scale between 0 and 100.
Efficiency of Composite Personalised Care (CPC) on clinical outcome (3) | at baseline, then 3 to 4 months and 6 to 8 months after the beginning of intervention
  - MADRS (Montgomery-Asberg depression scale). MADRS is a 10 -item scale that evaluates different aspects of depressive symptomatology. It provides a good estimation of the severity of depression and is sensitive to change.
Efficiency of Composite Personalised Care (CPC) on clinical outcome (4) | at baseline, then 3 to 4 months and 6 to 8 months after the beginning of intervention
  - Brief Psychiatric Rating Scale (BPRS). BPRS is a scale that evaluates general psychiatric symptomatology.
Efficiency of Composite Personalised Care (CPC) on clinical outcome (5) | at baseline, then 3 to 4 months and 6 to 8 months after the beginning of intervention
  PANSS (Positive and Negative Syndrome Scale) PANSS is a 30-item scale widely used in schizophrenia research to assess positive and negative psychotic dimensions as well as general symptomatology
Efficiency of Composite Personalised Care (CPC) on clinical outcome (6) | at baseline, then 3 to 4 months and 6 to 8 months after the beginning of intervention
  Clinical Global Impression (CGI) scale. CGI estimates the current severity, of illness on a 7-point scale, as well as evolution and therapeutic index in reference to the clinicians past experiences of similar patients (3 items).
Efficiency of Composite Personalised Care (CPC) on clinical outcome (7) | at baseline, then 3 to 4 months and 6 to 8 months after the beginning of intervention
  Clinical Global Impression (CGI) scale. CGI estimates the current severity, of illness on a 7-point scale, as well as evolution and therapeutic index in reference to the clinicians past experiences of similar patients (3 items).
Efficiency of Composite Personalised Care on linguistic and discourse markers | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  The recording of the interview will allow to extract reliable linguistic metrics that will be processed semi-automatically.
Efficiency of composite personalised care on neurological soft signs (1) | at baseline and 6 to 8 months after the beginning of intervention
  Neurological Soft Signs rating scale (NSS) assesses five factors: motor coordination, motor integration, sensory integration, quality of lateralization and involuntary movements or posture; as well as extrapyramidal symptoms (Simpson Angus Scale) and lateralization (Edinburgh questionnaire).
Efficiency of composite personalised care on neurological soft signs (2) | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Electronic Neurological Soft Signs (eNNS) This device incorporates a new, tablet-based and clinically suitable app (behavioral tasks), including tasks designed to probe balance of excitation/inhibition (multi-finger tapping task), body scheme tasks where finger posture recognition is measured and visuomotor sequence learning under variable cognitive load (using visual attentional distractors).
Efficiency of composite personalised care on cognitive complaints | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Subjective Scale to Investigate Cognition in Schizophrenia (SSTICS) is a 21-item Likert-type scale that allows a quantitative approach of cognitive complaint.
Efficiency of composite personalised care on cognitive functions (Verbal learning and memory) | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Hopkins Verbal Learning Test
Efficiency of composite personalised care on cognitive functions (Flexibility) | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  TMT A/B (Reitan, 1959)
Efficiency of composite personalised care on cognitive functions (Social cognition) | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Consensus autour de la COgnition Sociale (CLACOS) (PerSo)
Efficiency of composite personalised care on cognitive functions (Selective attention) | 3 to 4 Month and 6 to 8 Month after the beginning of intervention
  D2-R test
Efficiency of composite personalised care on cognitive functions (Verbal long-term memory) | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Hopskins Verbal Learning Test (HVLT) delayed recall
Efficiency of composite personalised care on cognitive functions (Visuospatial learning and memory) | 3 to 4 Month and 6 to 8 Month after the beginning of intervention
  Brief Visuospatial Memory test
Efficiency of composite personalised care on cognitive functions (Planning abilities) | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Shopping test (Martin 1972)
Efficiency of composite personalised care on cognitive functions (Speed processing) | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Wechsler Adult Intelligence Scale (WAIS) (code)
Efficiency of composite personalised care on cognitive functions (Inhibition control) | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Stroop (Incompatibility)
Efficiency of composite personalised care on cognitive functions (Visuospatial long-term memory) | 3 to 4 Month and 6 to 8 Month after the beginning of intervention
  Brief Visuospatial Memory test (BVMT) delayed recall
Efficiency of composite personalised care on cognitive functions (Working Memory) | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Wechsler Adult Intelligence Scale (WAIS) (Digit span)
Efficiency of composite personalised care on motivation | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Behavioral inhibition system (BIS) and behavioral activation system (BAS)
Embodiment ability in virtual reality environment | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Embodiment ability in virtual reality environment will be assessed using a simulation of two districts of a lively city via the Vive Pro virtual reality kit
Effect of Composite Personalised Care on Health-related quality-of-life (1) | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Short Form -12 items quality of life questionnaire (SF-12) SF-12 is a multipurpose self-report measure of both physical and mental health status
Effect of Composite Personalised Care on Health-related quality-of-life (2) | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  European Quality of Life - 5 Dimensions - 5 Levels (EQ-5D-5L)
  EQ-5D-5L investigates 5 dimensions: mobility, self care, usual activities, pain/discomfort, anxiety/depression. These 5 dimensions are rated on 5 levels ranging from no problems to extreme problems.
Effect of Composite Personalised Care on medication adherence | at baseline, 3 to 4 months and 6 to 8 months after the beginning of intervention
  Medication adherence (MARS) is a short assessement (5 items) of the adherence to medication
Acceptability of the program for the e-Health application | 3 to 4 months after the beginning of intervention
  amount of time spent on the application
Patient's satisfaction with the e-health application | 3 to 4 months after the beginning of intervention
  satisfaction score measured by the User Version of the Mobile Application Rating Scale (uMARS)
Level and changes of biological markers (metabolism of monocarbon compounds) | at baseline and 6 to 8 months after the beginning of intervention
  dosage of folates, B12 vitamin, homocysteine
Level and changes of biological markers (lipid membranes) | at baseline and 6 to 8 months after the beginning of intervention
  lipid composition of the red blood cells membrane, including the major lipid classes, such as phosphatidylcholine (PC), phosphatidylserine (PS), sphingomyelin (SM), phosphatidylethanolamine (PE), PE plasmalogen and their molecular species)
Longitudinal epigenetic and seric changes associated with outcome (1) | at baseline and 6 to 8 months after the beginning of intervention
  Levels of RNA (messenger RNA, microRNA, long non-coding RNA) will be assessed using next generation sequencing methods.
Longitudinal epigenetic and seric changes associated with outcome (2) | at baseline and 6 to 8 months after the beginning of intervention
  Levels of RNA (messenger RNA, microRNA, long non-coding RNA) will be assessed using next generation sequencing methods.
Cost-effectiveness of Composite Personalised Care | at the end of the follow-up, up to 4 years
  Incremental cost-effectiveness ratios (ICER) will assess the efficiency of CPC vs. TAU (overall and by component). They will be expressed in cost per quality-adjusted life-years (QALY) gained and in cost per PSP point gained.
Budgetary impact analysis of the generalization of Composite Personalised Care | at the end of the follow-up, up to 4 years
  Total costs and health benefits associated with generalizing CPC will be assessed and compared to TAU over a 5-year period.

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHRU Brest, Brest
  - Centre Esquirol - CHU CAEN, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Centre Hospitalier La Chartreuse, Dijon
  - Hôpital Fontan, Lille
  - Hôpital La Colombière - CHU Montpellier, Montpellier
  - Eldorado - Maison des Adolescents de Meurthe et Moselle, Nancy
  - CH Orsay, Orsay
  - GHU Paris Neurosciences Psychiatrie, Paris
  - Nineteen GHU, Paris
  - CHU Poitiers, Poitiers
  - C.H. Guillaume Regnier, Rennes
  - CHU Purpan, Toulouse